CLINICAL TRIAL: NCT06933082
Title: Efficacy of the Health Beliefs Model - Based Intervention in Enhancing Workers' Adherence to Wearing Personal Protective Equipment in Diyala State Company:
Brief Title: Health Beliefs Model, Enhancing Workers' Adherence,Personal Protective Equipment
Acronym: HBM PPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Nedaa Qahtan Touma, PhD. student, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1/3/1/8/3812 on 27 May 2024
Record Dates: First submitted 2025-04-03; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Occupational Toxicity and Health Hazards of the Healthcare Providers at Healthcare Facilities in Sulaimani City, Iraq

STUDY DESIGN:
Intervention Model Description: At first, all participants in both groups underwent a pre-test to provide them with basic data. Then, the researcher applied the educational Program to the study group only using group lectures, PowerPoint Presentations, Posters, illustrations, and group discussion sessions. The Program includes five lectures, each lasting 40 minutes. Each one focused on specific topics and objectives, where the focus was on what occupational hazards, types of occupational hazards, are and how to prevent these hazards in the work environment, and presenting some statistics that were previously conducted in the same company to make workers know more about these hazards and adopt healthy behavior to prevent them. A guide was provided to these participants at the end of the educational intervention. Two follow-up sessions were held after the end of the intervention Program and after two months. All training sessions were held in conference room in Diyala state company. There was no training for the contro
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- personal protective equipment (Experimental): The concept of perceived susceptibility: The worker's belief about the possibility of developing occupational hazards or accident.
  1. Explain the concept of occupational diseases or hazards.
  2. Present statistical studies on occupational hazards or diseases.
  3. Types of occupational hazards
  The second lecture includes:
  Perceived severity Concept: A worker's belief about the severity of occupational hazards or accident include explain the impact of these risks on the health of workers and infrastructure.
  A. Physical hazard effects. B. Psychosoical hazard effects. C. Chemical hazard effects. D. Mechanical hazard effects. E. electrical hazard effects F. Biological hazard effects. The concept of perceived barriers: the worker's belief about the effects that prevent him from preventing occupational hazards such as Contraindications for the use of personal protective equipment by the worker.
  Interventions: Behavioral: An intervention program has been developed acceding to The field visit conducted by researcher before the start of the study and observed the work environment and the lack of commitment of workers t

INTERVENTIONS:
Behavioral: An intervention program has been developed acceding to The field visit conducted by researcher before the start of the study and observed the work environment and the lack of commitment of workers t — An intervention program has been developed acceding to The field visit conducted by researcher before the start of the study and observed the work environment and the lack of commitment of workers to implementing the occupational health and safety program despite the existence of this program in the company.this intervention program based on health belief model in improventing workers' adherence related to occupatioan hazards prevention by wearing PPE. Validity and pre-test are applied prior to the implementation of the intervention program. The program is comprised of five main lecture each lecture is designed and scheduled for at least (45) minutes which deals with changing of workers' health beliefs about occupatioan hazards prevention.All lectures are presented at conference hall in the company.The implementation of health intervention program is initiated during the period of June 20th, 2024 to June 25th, 2024. Each lecture is designed and scheduled for approximately (45)

SUMMARY:
Personal protective equipment is designed to protect workers from serious workplace injuries or illnesses resulting from contact with chemical, radiological, physical, electrical, mechanical, or other workplace hazards. It may include items such as gloves, safety glasses and shoes, earplugs or muffs, hard hats, respirators, and full body suits.

True experimental design, using randomized controlled trial approach, is carried throughout the present study to determine the efficacy of applying the Health Beliefs Model in enhancing health behaviors of workers related to personal protective equipment wear at Diyala state company for the period of February 1 2024 through January 1 2025.

The sample of the study is A probability, simple random sample and it consist of (100) worker, who are work at factories in Diyala state company .The sample is randomly selected and assigned to the study and control groups of (50) workers each for who are equally distributed from each factory.

The intervention for the study group involved a health intervention lecture about occupational hazards and personal protective equipment used based on HBM. Analyzed data using SPSS, Version 23 using descriptive statistics, and inferential statistics and mixed design analysis of variance (ANOVA).

Findings of this study depict that there were statistically significant differences among all concepts of the HBM related to occupational hazards prevention by using PPE.

This study concluded that Applying HBM demonstrates the importance of PPE use in prevention of occupational hazard or accident in workplace and has a positive impact on workers' behaviors.

DETAILED DESCRIPTION:
Occupational Exposure to Lead, Nickel and Copper among Workers in Diyala State Company, The objective of this study was assessment occupational exposure to Pb, Ni, and Cu metals of workers in Diyala state company. Eighty two blood samples were collected (58 blood samples from workers working in the Diyala State Company and 24 samples from control samples for employees who don't relate with industrial emissions). Five ml. of venous blood was withdrawn for each sample. The concentration of Pb, Ni and Cu in the blood samples was determined by using the Flame less Atomic Absorption Spectrometer (FLAAS), depending on the years of work, high levels of Pb, Ni, and Cu in company workers than controls with significant differences (p<0.05). the investigates noticed increase levels of Pb, Ni, and Cu with occupation period progression, where it is found the levels of Pb, Ni, and Cu scored highest mean within 21-34 occupation period, and least mean value at <1 occupation period . Based on occupational places, investigates noticed highest levels of Pb in Iron heart worker , Ni level was highest in painting worker , and Cu level was highest in wires worker and least of all metals was at controls. Depending on age stages, investigates showed increase levels of Pb, Ni, and Cu with age stages progression, where it is found the levels of Pb, Ni, and Cu scored highest mean within >50 age stage, while the least mean value of Pb, and Cu at 3-40 years age stage, and least mean value of Ni was at <30 age. Finally, we notice there are positive correlations among metals and workers age.

ELIGIBILITY:
Inclusion Criteria:

* workers' working in factories with high occupational hazards and morning staff work.

Exclusion Criteria:

officials , administrative department employees,employees who did not agree to participate and those who are work in evening shift.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
The data were analyzed and interpreted through use of the application of Statistical Package for Social Sciences (SPSS), version 26.0. | Four weeks after administering the applied HBM Intervention (July 25th, 2024) the researcher performed posttest-I for all study participants. Then, eight weeks later (25 Septamber, 2024) the researcher performed posttest-II.
  The data were analyzed using the Statistical Package for Social Sciences (SPSS), version 26.0. Descriptive statistics, including mean and standard deviation, were calculated for the data. To explore group differences over time regarding wearing personal protective equipment to prevent or reduce occupational hazards, a repeated measures ANOVA was conducted. The Spear man correlation was used to examine the relationships between variables, while the point-bi-serial correlation was employed to find the association between binary and continuous variables. Normality of the data was tested using the Kolmogorov-Smirnov test.

CONTACTS AND LOCATIONS:
Locations (2):
- Iraq (2):
  - Iraqi/ Diyala state company, Baghdad
  - Diyala state company, Baqubah

REFERENCES:
- See also: Related Info — http://orcid.org/0009-0009-6928-7357